CLINICAL TRIAL: NCT02411279
Title: Anticipation and Detection of Heart Failure Decompensation With Automatic Treatment of Informations Derived From Non Intrusive Sensors and Devices
Brief Title: Anticipation and Detection of Heart Failure Decompensation With Automatic Treatment of Informations
Acronym: e-INCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6155
Record Dates: First submitted 2015-03-17; First posted 2015-04-08 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure
Keywords: Heart failure; telemonitoring; intrusive sensors; intrusive devices; Heart failure stage II; Heart failure stage III; heart disease
MeSH Terms: conditions — Heart Failure; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Groupe 1: experimental group: Equiped group with telemedicine systems
  Interventions: Other: Equiped group with telemedicine systems
- Groupe 2: control group: Non equiped group with telemedicine systems

INTERVENTIONS:
Other: Equiped group with telemedicine systems
  Groups: Groupe 1: experimental group

SUMMARY:
Heart failure (HF) is a serious chronic disease with frequent readmissions, some of which can be prevented by early action. The management of HF is complex: long, often difficult and costly. In France, nearly one million people suffer from HF and 120,000 new cases are diagnosed every year. With the aging population, this number will continue to evolve and become a real public health problem. Within 10 to 20 years ahead, WHO projects that heart failure in either the 3 most common diseases in industrialized countries.

The objective of the project is to test an intelligent platform for monitoring at home, using non-intrusive sensors, patients with heart failure, particularly those with stage II and III NYHA. It will assist the medical automating the processing of information from these sensors to detect and report an early stage risk situations.

Patient monitoring, by a system of telemedicine tools associated with motivation and education helps significantly reduce the number of days of hospitalization becomes important when the patient is hospitalized for acute HF.

ELIGIBILITY:
Inclusion Criteria:

* Population with heart failure stage II and III

Exclusion Criteria:

* Population whose age is less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with heart failure stage II and III
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Anticipation and detection of heart failure with automatic treatment of information derived from non intrusive sensors and devices | patient's medical data will be controlled remotely by health professional for the duration of hospital stay, up to 1 year]

CONTACTS AND LOCATIONS:
Overall Officials: ANDRES Emmanuel, MD, PhD, Principal Investigator — Strasbourg University Hospital, France
Locations (1):
- Service de Médecine Interne, diabète et maladies métaboliques - Médicale B, Strasbourg, France